CLINICAL TRIAL: NCT02145897
Title: A Prospective, Multicentric, Phase I/II, Open Label, Randomized, Interventional Study to Evaluate the Safety and Efficacy of Intramuscular and Intravenous Administration of Autologous ADMSCS for Treatment of Critical Limb Ischemia (CLI).
Brief Title: To Evaluate the Safety and Efficacy of IM and IV Administration of Autologous ADMSCs for Treatment of CLI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/CLI/11-12/001
Record Dates: First submitted 2014-05-08; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Critical Limb Ischemia
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologous Stromal Vascular Fraction (Experimental): single dose of autologous adipose derived Stromal Vascular Fraction (SVF) SVF divided in two fraction and infused intravenously and intramuscularly
  Interventions: Biological: Autologous Stromal Vascular Fraction (SVF)
- Autologous Adipose Derived MSCs (Experimental): One dose of 1 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intravenously and one dose of 1 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intramuscularly
  Interventions: Biological: Autologous Adipose Derieved MSCs
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Biological: Autologous Stromal Vascular Fraction (SVF) — Study arm A subjects will receive single dose of autologous adipose derived Stromal Vascular Fraction (SVF) SVF divided in two fraction and infused intravenously and intramuscularly
  Other Names: Autologous Stromal Vascular Fraction
  Arms: Autologous Stromal Vascular Fraction
Biological: Autologous Adipose Derieved MSCs — Study arm B subjects will receive one dose of 1 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intravenously and one dose of 1 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intramuscularly
  Arms: Autologous Adipose Derived MSCs
Other: Control
  Arms: Control

SUMMARY:
Various preclinical animal studies have shown the potential of stem cells in re-vascularising ischemic limbs and promoting collateral vessel formation. SVF have the potential to facilitate the formation of new blood vessels and skeletal muscle. Early pilot clinical studies indicate that stem-cell transplantation is feasible and may have beneficial effects in CLI. Injury or inflammation is a prerequisite for the participation of circulating stem cells to home and differentiate on to this microenvironment. The increased vascular permeability and expression of adhesion proteins like integrin assist in stem cell homing. The migratory capacity of stem cells is dependent on natural growth factors such as vascular endothelial growth factor (VEGF), Stromal cell derived factor (SDFI) and stem cell factor (SCF). The expression of VEGF, SDFI and SCF is highly unregulated in the hypoxic muscular tissue and is responsible for the recruitment of the stem cells to assist in the repair mechanism and consequent improvement in limb function.

In addition to the above regenerating potential of SVF, they have several advantages; they can be easily isolated without further culturing it. Most importantly SVF have shown to have significantly highest expression of pluripotent markers similar to that of human embryonic stem cells and yet they are non-tumorogenic and safe.

MSCs are having angiogenic activity and hence may be excellent source to develop neo-vasculature and hence could be explored for their therapeutic potential for treating Critical Limb Ischemia. MSC's also display membrane-bound and insoluble secreted molecules involved with cell attachment to neighbouring cells and to the extra cellular matrix19 Adipose derived Stromal vascular fraction and Mesenchymal Stem Cells has been found in preclinical studies to be safe and effective.

The current Phase I/II study of adipose derived stromal vascular fraction and Mesenchymal stem cells is conducted with the broad objective of establishing safety and efficacy.

DETAILED DESCRIPTION:
Adipose Derived Stromal Vascular Fraction (ADSVF) Stromal Vascular Fraction (SVF) obtained from tumescent liposuction. The SVF contains a variety of cells such as pre-adipocytes, endothelial cells, smooth muscle cells, pericytes, fibroblasts, and adult stem cells (ASCs). In addition, the SVF also contains blood cells from the capillaries supplying the fat cells. These include erythrocytes or red blood cells, B and T cells, macrophages, monocytes, mast cells, natural killer (NK) cells, hematopoietic stem cells and endothelial progenitor cells, to name a few. It also contains growth factors such as transforming growth factor beta (TGF-β), platelet-derived growth factor (PDGF), and fibroblast growth factor (FGF), among others. This is consistent with the secretions of cells in the presence of an extracellular matrix. The SVF also contains the various proteins present in the adipose tissue extracellular matrix of which laminin is of interest due to its ability to help in neural regeneration.Entire procedure for SVF preparation and isolation of SVF cells will be carried out in cGMP compliance clean room.

Pure stromal vascular fraction to the tune of 99% will be isolated for this clinical trial eliminating other unnecessary cells such as RBC and leukocytes.

Adipose Derived Mesenchymal Stem Cells (ADMSC) Human mesenchymal stem cells (MSCs) are present as a rare population of cells in adipose tissue which is almost 30-40% of the nucleated cells, but they can rapidly grow in culture without losing their stemness. MSCs can be expanded in vitro ≥ 2 million -fold and retain their ability to differentiate into several mesenchymal lineages. MSCs have several characteristics such as Ease of isolation, High expansion potential,Genetic stability,Reproducible attributes from isolate to isolate,Reproducible characteristics, Compatibility with tissue engineering principles, Potential to enhance repair in many vital tissues, Uniform dose and Better quality control and release criteria.

Beside autologous use MSC can also be used for allogenic therapy. Several studies have used allo-MSC in vivo and experience suggests that the allo-MSCs are not rejected and many have positive effects on engraftment.MSC's can be isolated from various tissues, cultured ex vivo, and expanded many fold.18 Cultured-expanded MSC's appear to represent a homogeneous population by flow cytometric measures of cell-surface markers. These cell retain the ability to undergo in vitro differentiation to osteogenic, adipogenic and chondrogenic lineages, even when clonally expanded.19 Human adipose tissue derived MSCs are capable of differentiating into endothelial cells in vitro and later form capillary-like structures in semisolid medium and suggest differentiation potential of MSCs is not restricted to mesodermal lineages but also transdifferentiation of MSCs into other lineages like endothelial could be realized in vitro and in vivo8 MSCs are known to give rise to limb-bud mesoderm (osteoblasts, chondrocytes, adipocytes, stroma cells, and skeletal myoblasts) and can also differentiate into cells of visceral mesoderm (endothelial cells).9 MSCs can facilitate vasculogenesis by increasing vascular endothelial growth factor (VEGF) levels. After MSCs are intramyocardially injected into the infarct zone, local VEGF levels rise, vascular density and regional blood flow increases, and contractility improves.

MSCs are having anti-fibrotic activity and hence may be excellent source to tackle pulmonary fibrosis and hence could be explored for their therapeutic potential for treating Idiopathic pulmonary fibrosis. MSC's also display membrane-bound and insoluble secreted molecules involved with cell attachment to neighboring cells and to the extra cellular matrix.18 This cell surface configuration may enable mesenchymal stem cells to home from bloodstream to mesenchymal tissue.

ELIGIBILITY:
Inclusion Criteria:

* 1. Critical limb ischemia (rest pain, un-healing wound/ulcer lasting more than 4 weeks)

  2. Category 4 & 5 Rutherford-Becker peripheral vascular disease affecting at least one limb with or without un-healing ulcer/wound of grade I or II on the Wagner scale

  3. Ankle -brachial index <0.6

  4. TcpO2 < 45 mm Hg measured at toe

  5. Life expectancy more than 2 years

  6. Subjects (male and female), aged 18 to 65 years (both inclusive)

  7. Glycosylated hemoglobin (HbA1C) ≤7 %

  8. INR value of below 2 before liposuction procedure

  9. Subject should be compliant to the treatment regimen follow like insulin, anti-diabetic drugs for the entire duration of the clinical study

  10. Subject who are not currently on or have discontinued treatment with immune-suppressants and/or corticosteroids within at least 20 days prior to screening

  11. Subject willing to give Informed Consent

Exclusion Criteria:

1. Uncontrolled high blood pressure
2. Uncontrolled diabetes with Glycosylated hemoglobin (HbA1C) > 7%
3. Severe cardiac insufficiency (Ejection fraction < 35%)
4. Frank infected ulcers with purulent discharge resulting in excessive infections, ulcers with exposed bone, fascia, joints, ligaments or tendons (Category 6 Rutherford-Becker peripheral vascular disease)
5. Subject diagnosed with cancer undergoing chemotherapy.
6. Poor nutritional status as measured by serum albumin <3.0 g/dL.
7. Severe anemia Hb < 7g/dl.
8. Subject had a leg revascularization surgery or history of amputation within the last 6 months or be a candidate for revascularization surgery during the course of the study.
9. Other unusual or rare forms of diabetes mellitus, or history of diabetic ketoacidosis or osteomyletis.
10. Subject unfit to undergo lipoaspiration as determined by the surgeon.
11. Subject has a history of bleeding disorder or clotting disorder
12. Have any condition, disease, disorder, or clinically significant laboratory abnormality that, in the opinion of the Investigator, would jeopardize the subjects' appropriate participation in this study or obscure the effects of treatment.
13. Pregnant or lactating women or women of child-bearing potential not using medically acceptable methods of contraception or women with positive urine pregnancy test (UPT) at screening
14. Subjects unwilling or unable to comply with the study procedures
15. Have received treatment with any investigational product (IP) or participated in any investigational study within 30 days or 5 half-lives of the IP, whichever is longer, before the Screening Visit.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
To assess the safety | 9 months
  The Incidence of treatment emergent Adverse Event (AE) in the study.

SECONDARY OUTCOMES:
To assess the efficacy | 9 months
  To explore the efficacy by assessing the potential of autologous adipose derived stromal vascular fraction and ex vivo expanded mesenchymal stem cells in alleviating the symptom of Critical Limb Ischemia (CLI)

OTHER OUTCOMES:
Safety | 9 months
  The safety parameters are composite of the following measures- Assessment of clinical laboratory parameters Assessment of vital signs Assessment of electrocardiogram (ECG) parameters
Efficacy | 9 months
  The efficacy parameters are composite of the following measures-
  1. Change in Transcutaneous oxygen pressure
  2. Change in Ankle brachial index (ABI)
  3. Change in the number of debridements in the study group as compared to the control group.
  4. Changes in wound cover changes in the study group as compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Arun B Bal, M.B.B.S.M.S., Principal Investigator — SL Raheja Hospital; Dr. Ashish S Johari, M.B.B.S.M.S., Principal Investigator — Jaslok Hospital and Research Centre; Dr. Meena Kumar, M.B.B.S.M.S., Principal Investigator — L T M C and L T M M General Hospital ,Sion; R Shekhar, M.B.B.S.M.S., Principal Investigator — Kokilaben Dhirubai Ambani Hospital and Medical Research Institute
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India